CLINICAL TRIAL: NCT06990958
Title: Erector Spinae Plane Block Versus Fascia Iliaca Compartment Block for Analgesia in Proximal and Midshaft Femur Surgeries in Adult Patients: A Randomized Controlled Study
Brief Title: Comparing Erector Spinae and Fascia Iliaca Blocks for Pain Relief After Femur Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Wissam Ahmed Mohamed El Damacey, Lecturer of Anesthesia, surgical ICU and Pain Management Faculty of Medicine, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MS-212-2023
Record Dates: First submitted 2025-05-18; First posted 2025-05-25 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Analgesia After Fracture Femur Surgeries
Keywords: Fascia iliac block, erector spinae block, femur fracture, adult analgesia
MeSH Terms: conditions — Femoral Fractures; Agnosia | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESPB Group (Active Comparator): patients was placed in the lateral position . the block was performed bz ipsilateral injection of a mixture containing 15mls bupivcaine 0,5% and 20mls normal saline.
  Interventions: Procedure: Erector Spinae Plane Block (ESPB) group
- FICB (Active Comparator): Patients was placed insupine position . the block performed using a mixture of 15mls bupivcaine 0,5% and 20mls normal saline.
  Interventions: Procedure: Fascia iliaca compartment block (FICB)

INTERVENTIONS:
Procedure: Erector Spinae Plane Block (ESPB) group — ultrasound guided erector spinae plane block (at lumbar level) in lateral position .
  Arms: ESPB Group
Procedure: Fascia iliaca compartment block (FICB) — ultrasound guided suprainguinal approach in supine position
  Arms: FICB

SUMMARY:
This clinical study compares two types of nerve blocks used to control pain in adult patients undergoing surgery on the upper (proximal) or middle (midshaft) part of the femur (thigh bone). The two blocks being studied are the Erector Spinae Plane (ESP) block and the Fascia Iliaca Compartment (FIC) block. Both techniques are commonly used in hospitals to reduce postoperative pain.

The goal is to determine which nerve block provides more effective pain relief, reduces the need for opioid medications, and supports faster recovery in patients following femur surgery. Results from this study may improve pain management strategies for similar procedures in the future.

Adults scheduled for proximal or midshaft femur surgery may be eligible to participate. Eligibility is determined based on clinical criteria reviewed by the study team.Administration of one of the two nerve blocks before surgery.Standard surgical and postoperative care.

Monitoring of pain levels at specific time points after surgery

Recording of opioid medication usage

Evaluation of patient satisfaction and any side effects related to the nerve block

Duration:

The intervention (nerve block) is administered once before surgery. Data collection continues during the immediate postoperative period and for a short time following surgery to assess outcomes.

Both nerve blocks are considered safe and are regularly used in clinical practice.

All procedures are performed by qualified clinicians, and safety monitoring is conducted throughout the study.

Participants may experience improved pain relief and reduced need for opioid medications. While direct benefit cannot be guaranteed, information gained from the study may help improve pain management for future patients undergoing similar surgeries.

Participation in the study is completely voluntary. Patients may choose not to participate or may withdraw from the study at any time without affecting the quality of their medical care.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80
* American society of Anathesiologist physical status ASA Ior II
* Patients undergoing Fixation of femur fractures

Exclusion Criteria:

1. Refusal of participation in study.
2. Bleeding disorders (platelets count < 80,000, INR >1.5, Prothrombin concentration < 60%).
3. Skin lesion, wounds or infection at the puncture site. Known allergy to local anesthetic drugs.
4. Known local anesthetic (LA) drug sensitivity. -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2025-03-05 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
duration of the block | 15 minutes after extubation till 24 hours postoperative
  time starting immediatelyafter giving the block till the first postoperative analgesic rescue which will be used if the pain score exceeds 4/10

CONTACTS AND LOCATIONS:
Locations (1):
- kasr alainy hospital -Cairo university , cairo, Cairo, Egypt